CLINICAL TRIAL: NCT04621825
Title: Post Market Surveillance Study to Confirm the Safety and Performance of the Silicone Subcategory of PHMB Foam Dressings in Chronic and Acute Wounds
Brief Title: Post Market Surveillance Study to Confirm Safety and Performance of Silicone PHMB Foam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: Imarc Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHMB Silicone 001
Record Dates: First submitted 2020-10-13; First posted 2020-11-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-01

CONDITIONS: Wound
Keywords: Antimicrobial PHMB; Silicone Foam; Chronic Wounds; Acute Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned intervention (Experimental): ActivHeal Silicone PHMB Adhesive and Non Adhesive Foam.
  Subjects will undergo treatment of their chronic or acute wound as indicated in the instructions for use with ActivHeal Silicone PHMB Adhesive and Non Adhesive Foam.
  Interventions: Device: ActivHeal Silicone PHMB Foam Adhesive and Non Adhesive dressing.

INTERVENTIONS:
Device: ActivHeal Silicone PHMB Foam Adhesive and Non Adhesive dressing. — Assigned interventions Subjects will undergo treatment of their chronic and acute wounds as indicated in instructions for use with ActivHeal Silicone PHMB Foam adhesive and Non Adhesive Foam dressings.
  Subjects will be evaluated as follows:
  Full Patient and wound assessment, Informed consent. Wound Assessment, application of dressings, (At each scheduled dressing change.) Wound Assessment, removal of dressings, (At each scheduled dressing change.) The patients will be evaluated at each dressing change over a four - six-week period (per AMS Product) or until the wound is healed to extent that the use of the ActivHeal Silicone PHMB Foam adhesive and Non Adhesive Foam dressings. is no longer indicated from the time that the patient has been recruited.
  The assessment of the presence and reduction of the signs and symptoms of Infection.

SUMMARY:
Post market surveillance study to confirm the safety and performance of Silicone Subcategory of PHMB Foam Dressings in Chronic and Acute Wounds.

DETAILED DESCRIPTION:
The design of the study is an open label, multicentre, single arm trial with subjects with moderate to heavily exuding chronic and acute wounds consisting of pressure ulcers, leg ulcers, diabetic leg and foot ulcers, surgical wounds first degree superficial and partial thickness burns. The performance data from this study will support clinically meaningful rates of successful improvement in the signs and symptoms of infection, without refection during 6- week treatment and follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Have a pressure ulcer, leg ulcer, diabetic leg and foot ulcer, surgical wound, first degree superficial burns or partial thickness second degree burns that are infected following assessment of signs and symptoms of infection with moderate to heavy levels of exudate.
* Have wounds at high risk of infection.
* Males or females, age 18 years or above.
* Subjects who are able to understand and give informed consent to take part in the study.

Exclusion Criteria:

* Subjects who are known to be non compliant with medical treatment.
* Subjects who are known to be sensitive to any of the device components, known sensitivity to PHMB.
* Subject is pregnant or actively breastfeeding.
* Subject has any significant or unstable medical or psychiatric condition, that in the opinion of the investigator, would interfere with his/her ability to participate in the study.
* Subject is currently in another clinical study.
* Patients who have a current illness or condition, or who have had an illness in the last 30 days which in the opinion of the investigator may interfere with wound healing (e.g. carcinoma, connective tissue disease, autoimmune disease or alcohol or drug abuse).
* Life expectancy of <6 months.
* Maximum burn area of >20% total body area in adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Effectiveness (performance) of the ActivHeal Silicone PHMB will be evaluated for efficacy success according to the following success criteria:
  Reduction in signs and symptoms of infection from baseline as defined as
  * The change from the Investigator's opinion of infection being present to no longer being present, or
  * If the Investigator determines infection is still present there is improvement in severity of at least two.
  No worsening of any signs/ symptoms of infection at 6 weeks or if infection resolved prior to 6 weeks, that no new evidence of infection occurred during the 6 week treatment follow up.

SECONDARY OUTCOMES:
Safety of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing. | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Safety will evaluated as incidence of device related adverse events.
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing in terms of wound progression | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Wound progression, assessed as the change from baseline to end of follow up. Monitoring of tissue types %,decrease in devitalised tissue, size and depth of wound.
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing in terms of pain. | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Change in patient pain will be assessed using Visual Analogue Scale, VAS, from baseline to end of follow up. Pain will assessed by completion of a Visual Analogue Scale VAS (0= no pain to 10 = worst pain imaginable).
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing in terms of pain at dressing removal. | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Patient pain will be assessed on removal of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing. Pain will assessed by completion of a Visual Analogue Scale, VAS(0= no pain to 10 = worst pain imaginable).
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing in terms of peri wound skin. | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Changes in the peri wound skin, prevents maceration. (Allows the uptake of exudate into the dressing.) Relative score will be used to score maceration of zero (no maceration), one (minimal maceration), two (moderate maceration), and three (excessive maceration and need to withdraw patient from study). Success will be determined that over the evaluation an increased score would represent peri wound deterioration.
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing in terms of dressing removal. | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Did the dressing cause trauma on removal to the wound (prevents formulation of granulation tissue growth into the pores of the dressing). Clinician and patient satisfaction with the device (ease of removal and no pain or trauma on removal) will be assessed using a likert type scale. (Very satisfied, Satisfied and not Satisfied).
Effectiveness of the ActivHeal Silicone PHMB foam adhesive and Non Adhesive foam dressing in terms of repositioning. | Immediately following initial assessment, dressing removal every 7 days follow up visits, for 6 weeks.
  Can the dressing be repositioned and or lifted, securely placed back down. Clinician satisfaction with the device (conformability & ease of use) will be assessed using a Likert type scale. (Very satisfied, Satisfied and not Satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Thirumani Govender, MD, Principal Investigator — TASK Clinical Research Centre 1 Smal Street Bellville, 7530
Locations (3):
- South Africa (3):
  - Dr Thirumani Govender, Bellville, Cape Town
  - Delft Day Hospital Premises, Delft S., Cape Town
  - Brooklyn Chest Hospital, Ysterplaat, Cape Town